CLINICAL TRIAL: NCT01584739
Title: A Phase I, Single Centre, Double-Blind, Randomised, Placebo- Controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Inhaled Doses of AZD8683 in Healthy Volunteers and COPD Patients
Brief Title: AZD8683 Multiple Dose Study in Healthy Volunteers and Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D1883C00002; Eudract 2011-005588-25
Record Dates: First submitted 2012-04-02; First posted 2012-04-25 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: Safety; tolerability; healthy; COPD (chronic obstructive pulmonary disease); pharmacokinetic; pharmacodynamic; inhaled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD8683 (Experimental)
  Interventions: Drug: AZD8683
- Placebo to AZD8683 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8683 — Multiple dose, oral inhalation (Healthy volunteers) Multiple dose, oral inhalation (COPD patients)
  Arms: AZD8683
Drug: Placebo — Multiple dose, oral inhalation (Healthy volunteers) Multiple dose, oral inhalation (COPD patients
  Arms: Placebo to AZD8683

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending inhaled doses of AZD8683 in Healthy volunteers and repeated inhalation of one dose level of AZD8683 in patients with chronic obstructive pulmonary disease given once daily.

DETAILED DESCRIPTION:
A Phase I, Single Centre, Double-Blind, Randomised, Placebo- controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Inhaled Doses of AZD8683 in Healthy Volunteers and COPD patients

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers and healthy female volunteers of non-child bearing potential, aged 18 to 45 years inclusive with suitable veins for cannulation or repeated venepuncture - Healthy volunteers
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg inclusive - Healthy volunteers and COPD patients
* Be able to inhale from the Turbuhaler® inhaler according to given instructions as well as be able to perform spirometry -Healthy volunteers and COPD patients.
* Male COPD patients or female COPD patients of non-childbearing potential (post menopausal or surgically sterilised) aged ≥40 years at Visit 1 - COPD patients
* Female healthy volunteers and female patients ≤60 years must have a negative pregnancy test at screening and on admission to the unit - Healthy volunteers and COPD patients

Exclusion Criteria:

* Prolonged QTcF >450 ms or shortened QTcF <340 ms or family history of long QT syndrome - Healthy volunteers and COPD patients
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8683 or excipients:Healthy volunteers and COPD patients
* History or presence of gastrointestinal, pulmonary, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs - Healthy volunteers and COPD patients
* Any clinically significant illness (other than COPD), medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product - COPD patients
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product - Healthy volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety profile in terms of: adverse events, Supine vital signs (blood pressure and pulse rate), body temperature, ECG, Physical examinations, Laboratory variables (clinical chemistry, haematology and urinalysis), Spirometry | Up to 13 days post dose.
  No formal statistical tests will be performed

SECONDARY OUTCOMES:
AZD8683 single dose pharmacokinetics from blood and urine in healthy volunteers. | Blood: From days 1 and 15 - Pre-dose, 5, 15 and 30mons, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 hrs (also 96 and 120hrs and follow-up). Urine: From days 1 and 15: pre-dose and 6, 12, 24, 48 and 72hrs.
  PK parameters:Cmax; tmax -Time to max plasma concentration; t½ λz,AUC-Area under the plasma concentration time curve from zero to infinity;AUC(0-t)-Area under plasma concentration time curve from zero to time of the last measurable concentration; AUC(0-24);AUC(0-72)-Area under the plasma concentration-time curve from zero to 72 hours; CL/F; Vz/F-Apparent volume of distribution during terminal phase; MRT-Mean residence time; Ae; Ae(0-t)-Cumulative amount of AZD8683 excreted unchanged in urine from zero (predose) to time t; fe-Fraction of dose excreted unchanged in urine; CLR-Renal clearance.
AZD8683 multiple dose pharmacokinetics from blood and urine in healthy volunteers. | Blood: From days 1 and 15 - Pre-dose, 5, 15 and 30mins, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 hrs (also 96 and 120hrs and follow-up). Urine: From days 1 and 15: pre-dose and 6, 12, 24, 48 and 72hrs.
  PK paramaters:Cmax and Cmin (max and min plasma concentration);tmax;t½ λz-Terminal half-life; AUC(0-τ)-Area under the plasma concentration-time curve during the dosing interval; Cav-Average plasma concentration;CL/F-Apparent plasma clearance; Rac AUC(0-τ)-Accumulation ratio of AUC(0-τ)compared to AUC(0-24)Day1;Rac Cmax-Accumulation ratio of Cmax compared to Cmax Day 1;Ae(t1-t2), Ae(0-τ)-Amount of drug excreted unchanged in urine in a collection interval; and to the end of the dosing interval respectively;fe(0-τ)-fraction of drug excreted unchanged in urine during a dosing interva;CLR.
Description of the pharmacodynamic (PD) effects of AZD8683 in healthy volunteers in terms of : FEV1 and FVC. | Predose, 5mins, 30mins, 1hr, 2hrs, and 4hrs on days 1 and 15.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax).FEV = Forced Expiratory Volume in 1 second. FVC = Forced Vital Capacity.
Description of the pharmacodynamic (PD) effects of AZD8683 in COPD patients in terms of : FEV1 and FVC. | Predose, 5mins, 30mins, 1hr, 2hrs and 4hrs on days 1 and 12.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax).FEV = Forced Expiratory Volume in 1 second. FVC = Forced Vital Capacity.
Description of the pharmacodynamic (PD) effects of AZD8683 in healthy volunteers in terms of : supine blood pressures and pulse rate. | Pre-dose, 30mins, 60mins, 90 mins, 2hrs and 4hrs, on days 1 and 15.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax). For diastolic blood pressure the minimum value(Emin), will be used.
Description of the pharmacodynamic (PD) effects of AZD8683 in COPD patients in terms of : supine blood pressures and pulse rate. | Pre-dose, 30mins, 60mins, 90 mins, 2hrs and 4hrs on days 1 and 12.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax). For diastolic blood pressure the minimum value(Emin), will be used.
Description of the pharmacodynamic (PD) effects of AZD8683 in healthy volunteers in terms of : QT interval corrected for heart rate using Fridericia's formula and heart rate. | 30mins pre-dose and 25 mins, 5mins, 1hr 25 mins, 1hr 55 mins and 3 hr 55 mins, on days 1 and 15.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax).
Description of the pharmacodynamic (PD) effects of AZD8683 in COPD patients in terms of : QT interval corrected for heart rate using Fridericia's formula and heart rate. | 30mins pre-dose and 25 mins, 5mins, 1hr 25 mins, 1hr 55 mins and 3 hr 55 mins on days 1 and 12.
  Average effect over the first 4 hrs (Eav, AUEC(0-4)/4 hours).Peak effect during the first 4 hrs (Emax).

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, Study Director — AstraZeneca Research and Development SE-431 83 Molndal Sweden
Locations (1):
- London, United Kingdom